CLINICAL TRIAL: NCT07082231
Title: Cohort of Patients With Ulcerative Colitis or Polyps Followed in CHU de Bordeaux Associated With a Biocollection - COLIBRI
Acronym: COLIBRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/61
Record Dates: First submitted 2025-03-12; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease (IBD); Acute Severe Ulcerative Colitis
Keywords: Acute severe ulcerative colitis; Ulcerative colitis; Inflammatory bowel disease; Biobank
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulcerative Colitis Group (Active Comparator)
  Interventions: Other: Blood sample; Procedure: biopsy
- Non-Ulcerative Colitis with Polyps Group (Placebo Comparator)
  Interventions: Other: Blood sample; Procedure: biopsy

INTERVENTIONS:
Other: Blood sample — 3 blood samples
Procedure: biopsy — 3 pairs of biopsy realised during the coloscopy

SUMMARY:
Ulcerative colitis (UC) is a chronic disease characterized by acute episodes of bloody diarrhea with varying degrees of severity. The most feared event, acute severe UC, can lead to life-threatening and systemic complications. Little is known about the determinants of severity in UC. The investigators hypothesize that distinct severity phenotypes of UC arise from intricated host-microbiota mechanisms influencing repair mechanisms. Our first and main objective is to study the natural history of UC during a one-year time period in a cohort of patients.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease characterized by acute episodes of varying-severity bloody diarrhea. Acute severe colitis poses systemic risks. In our pilot ITAC project, the investigators found a direct link between deep colonic ulcers and systemic inflammation in acute severe colitis, suggesting repair failure. Conversely, excessive repair in UC can lead to colorectal neoplasia, especially sessile serrated adenomas in remission cases.. The investigators plan to prospectively collect tissue and blood samples of patients with UC or non-UC patients with polyps undergoing endoscopy in the Gastroenterology unit or colectomy in the Abdominal surgery unit of CHU de Bordeaux. For all patients, additional biopsies will be collected for histology, microbiota characterization, transcriptomic profiling and cells phenotyping. Additional blood samples will be collected for immune cells phenotyping, genetic profiling, and multiplex cytokines measurement. Routine clinical, endoscopic and biological data will be collected using the Entrepot de Données de Santé of CHU de Bordeaux. The patients will be divided in groups based on the endoscopy phenotype: unactive disease, non-severe active disease, severe disease and on the presence of polyps. Patients without ulcerative colitis with polyps will be studied as a control group.clinical, endoscopic and biological data will be collected using the Entrepot de Données de Santé of CHU de Bordeaux. The patients will be divided in groups based on the endoscopy phenotype: unactive disease, non-severe active disease, severe disease and on the presence of polyps. Patients without ulcerative colitis with polyps will be studied as a control group.

ELIGIBILITY:
* Inclusion criteria:

  * General Inclusion Criteria:

    * Patients covered by a social security system.
    * French-speaking patients.
    * Patients aged ≥18 years.
    * Patients who have provided free, informed, and written consent (no later than the inclusion day and before any research-related examination).
  * Specific Inclusion Criteria for the UC Group:

    * Patients diagnosed with ulcerative colitis (UC) according to the European Crohn's and Colitis Organisation (ECCO) guidelines.
    * Patients undergoing lower gastrointestinal endoscopy or rectocolic surgery.
  * Non-UC Patients with Polyps Group:

    * Patients undergoing colonoscopy with resection of hyperplastic polyps in the rectum, sessile serrated lesions, or adenomas >2 cm.
* Exclusion criteria:

  * Patients with perianal, ileal lesions, or endoscopic features of colonic lesions suggestive of Crohn's disease.
  * Pregnant or breastfeeding women.
  * Patients under legal protection or unable to provide informed consent.
  * Patients deprived of liberty by judicial or administrative decision, hospitalized without consent, or admitted to a healthcare or social institution for reasons unrelated to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mayo clinical activity score | Baseline, Month 12
  Evolution of Mayo clinical activity score between inclusion and last visit. There is 4 items and for each item is rated from 0 to 3 and total score that varies from 0 to 12
UCEIS endoscopic activity score | Baseline, Month 12
  Evolution of UCEIS endoscopic activity score between inclusion and last visit. There is 3 items. Each item is rated from 0 to 2 or 0 to 3 and total score that varies from 0 to 8
Nancy histological activity score | Baseline, Month 12
  Evolution of Nancy histological activity score between inclusion and last visit.
  The Nancy index is defined by a 5-level classification ranging from grade 0 (absence of significant histological disease activity) to grade 4 (severely active disease).
Advanced therapy (biologics or small molecules) | Baseline, Month 12
  Number of new advanced therapy (biologics or small molecules) between inclusion visit and last visit
Hospitalization due to disease flare | Baseline, Month 12
  Number of hospitalization due to disease flare between inclusion visit and last visit
Colectomy | Baseline, Month 12
  Number of colectomy between inclusion and last visit

CONTACTS AND LOCATIONS:
Overall Officials: Pauline RIVIERE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No